CLINICAL TRIAL: NCT00976508
Title: Phase 1 Safety And Tolerability Study Of Figitumumab Combined With Pegvisomant In Patients With Advanced Solid Tumors
Brief Title: Figitumumab Combined With Pegvisomant For Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021040
Record Dates: First submitted 2009-09-10; First posted 2009-09-14 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Sarcoma
Keywords: advanced solid tumors cancer refractory cancer figitumumab pegvisomant
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Sarcoma | interventions — figitumumab; pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: figitumumab; Drug: pegvisomant

INTERVENTIONS:
Drug: figitumumab — IGF-1R antibody, 20 mg/kg, IV every 3 weeks for up to 1 year
  Other Names: CP-751,871
Drug: pegvisomant — growth hormone antagonist, 10, 20 or 30 mg per day via subcutaneous injection for up to 1 year
  Other Names: Somavert

SUMMARY:
This is a Phase 1 study investigating the safety and tolerability of Figitumumab plus Pegvisomant for treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This study was closed to enrollment on 18 April 2011 due to inability to recruit patients on a timely basis as well as business reasons. Study closure was not related to any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with advanced solid tumors for which the combination of figitumumab and pegvisomant are reasonable treatment options.
* Patients between the ages of 10 and 18 years with advanced sarcomas for which there is no available curative therapy or therapy proven to prolong survival with an acceptable quality of life will be included in the Sarcoma Expansion Cohort.
* Adequate recovery from prior therapies.
* Adequate organ function (i.e. bone marrow, kidney, liver)
* Total IGF-1 ≥100 ng/ml (13 nmol/L).

Exclusion Criteria:

* Concurrent treatment with any anti-tumor agents.
* Pregnant or breastfeeding females.
* Significant past history or active cardiac disease
* Active infection
* History of diabetes mellitus.
* Glycosylated hemoglobin >5.7

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (2):
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
- Pfizer Investigational Site, Montreal, Quebec, Canada
- Pfizer Investigational Site, Helsinki, Finland
- Pfizer Investigational Site, Münster, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021040&StudyName=Figitumumab%20Combined%20With%20Pegvisomant%20For%20Advanced%20Solid%20Tumors%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab 20mg/kg + Pegvisomant 10 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles, up to a maximum of 17 cycles (corresponding to 1 year). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 10 mg subcutaneously once daily, up to a maximum of 17 cycles (corresponding to 1 year). Each cycle was of 21 days.
- Figitumumab 20mg/kg + Pegvisomant 20 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles, up to a maximum of 17 cycles (corresponding to 1 year). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 20 mg subcutaneously once daily, up to a maximum of 17 cycles (corresponding to 1 year). Each cycle was of 21 days.
Period: Overall Study
Arm/Group | Figitumumab 20mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Started | 17 (18 subjects were enrolled; 17 subjects were treated; 1 subject was not eligible.) | 6
Completed | 3 (These subjects withdrew from last study treatment due to progressive disease.) | 0
Not Completed | 14 | 6
Not completed — Death | 7 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease Progression | 4 | 4
Not completed — Subject Enrolled in Hospice | 1 | 0
Not completed — Terminated by the Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Figitumumab 20 mg/kg +Pegvisomant 10 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles, up to a maximum of 17 cycles (corresponding to 1 year). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 10 mg subcutaneously once daily, up to a maximum of 17 cycles (corresponding to 1 year). Each cycle was of 21 days.
- Figitumumab 20 mg/kg + Pegvisomant 20 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles, up to a maximum of 17 cycles (corresponding to 1 year). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 20 mg subcutaneously once daily, up to a maximum of 17 cycles (corresponding to 1 year). Each cycle was of 21 days.
- Total: Total of all reporting groups
Arm/Group | Figitumumab 20 mg/kg +Pegvisomant 10 mg | Figitumumab 20 mg/kg + Pegvisomant 20 mg | Total
Number analyzed (Participants) | 17 | 6 | 23
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (17.4) | 32.3 (9.8) | 45.0 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. AEs were graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 (Grade [Gr] 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death). Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: From Screening to the follow-up visit (90 days after last dose of figitimumab)
Population: Safety analysis set: all enrolled participants who received at least 1 dose of either of the study medications.
Measure: Number; unit: Participants
Groups:
- Figitumumab 20mg/kg + Pegvisomant 20 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles, up to a maximum of 17 cycles (corresponding to 1 year). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 20 mg subcutaneously once daily up to a maximum of 17 cycles (corresponding to 1 year). Each cycle was of 21 days.
Arm/Group | Figitumumab 20mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 17 | 6
Participants
  Number of participants with AEs | 17 | 6
  Number of participants with SAEs | 9 | 4
  Number of participants with Gr 3 or Gr 4 AEs | 12 | 4
  Number of participants with Gr 5 AEs | 7 | 1

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLT was defined as any of the following events occurring during DLT period and considered related to study medication: Grade (Gr) 4 neutropenia lasting >=7 days, febrile neutropenia (Gr 3 or 4 neutropenia, fever >=38.5 degrees Celsius, lasting over 24 hours), neutropenic infection (Gr >=3 neutropenia, infection); Gr 3 or 4 thrombocytopenia associated with bleeding or Gr 4 thrombocytopenia >=7 days; Gr 3 or 4 lymphopeniab accompanied by an opportunistic infection; other non-hematologic Grade 4 toxicities or symptomatic Gr 3 toxicities that require medical intervention and 14 days to resolve.
Time Frame: From Cycle 2, Day 1 to Cycle 3, Day 8; from Cycle 1, Day 15 to end of Cycle 2
Population: Safety analysis set: all enrolled participants who received at least 1 dose of either of the study medications. N=number of participants remained on treatment throughout the required DLT period and included as analyzed for DLT based on the defined DLT evaluability specifications.
Measure: Number; unit: participants
Groups:
- Figitumumab 20 mg/kg + Pegvisomant 10 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles, up to a maximum of 17 cycles (corresponding to 1 year). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 10 mg subcutaneously once daily up to a maximum of 17 cycles (corresponding to 1 year). Each cycle was of 21 days.
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 6 | 6
participants | 1 | 0

3. Secondary Outcome: Serum Circulating Insulin-like Growth Factor (IGF-1) Levels
Description: The effect of the combined therapy with figitumumab and pegvisomant on circulating concentrations of total IGF-1 was assessed.
Time Frame: Days 1 and 15 of Cycle 1 (Baseline); Day 1 of subsequent cycles starting from Cycle 2 to Cycle 27; end of treatment (21 days after last dose of figitumumab); follow-up visit (90 days after last dose of figitumumab)
Population: Biomarker analysis set: all enrolled participants who had at least 1 baseline or on-study sample submitted. N=number of participants who were evaluable for IGF-1 Levels at prespecified time points.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 17 | 6
nanogram/milliliter (ng/mL)
  Baseline/Cycle 1 (n = 16, 6) | 150.18 (77.06) | 189.17 (59.79)
  Cycle 2 (n = 12, 6) | 725.72 (497.12) | 498.50 (218.28)
  Cycle 3 (n = 6, 5) | 474.53 (418.39) | 247.40 (147.41)
  Cycle 4 (n = 5, 3) | 542.09 (510.84) | 124.67 (83.94)
  Cycle 5 (n = 3, 4) | 990.40 (542.21) | 248.25 (127.43)
  Cycle 6 (n = 2, 2) | 1369.5 (161.93) | 122.50 (137.89)
  Cycle 7 (n = 1, 2) | 1594.00 (NA) — The data was not analyzed since only 1 out of 17 participants were evaluable at this time-point. | 272.50 (105.36)
  Cycle 8 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 501.00 (94.75)
  Cycle 9 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 331.00 (229.10)
  Cycle 10 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 412.50 (185.97)
  Cycle 11 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 426.50 (119.50)
  Cycle 12 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 375.50 (350.02)
  Cycle 13 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 457.50 (36.06)
  Cycle 14 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 420.00 (45.25)
  Cycle 15 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 444.50 (47.38)
  Cycle 16 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 443.50 (23.33)
  Cycle 17 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 426.00 (4.24)
  Cycle 18 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 570.50 (487.20)
  Cycle 19 (n = 0, 1) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 537.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.
  Cycle 20 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 458.50 (239.71)
  Cycle 21 (n = 0, 2) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 437.00 (21.21)
  Cycle 22 (n = 0, 1) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 401.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.
  Cycle 23 (n = 0, 1) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 481.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.
  Cycle 24 (n = 0, 1) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 361.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.
  Cycle 25 (n = 0, 1) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 424.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.
  Cycle 26 (n = 0, 1) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | 366.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.
  Cycle 27 (n = 0, 0) | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point. | NA (NA) — The data was not analyzed since no participants were evaluable at this time-point.
  Follow-Up (n = 2, 1) | 791.50 (813.88) | 1285.00 (NA) — The data was not analyzed since only 1 out of 6 participants were evaluable at this time-point.

4. Secondary Outcome: Cycle 1: Maximum Observed Plasma Concentration (Cmax) of Figitumumab
Time Frame: Cycle 1: Day 1 (within 2 hours before figitumumab infusion), Day 2 (1 hour post figitumumab infusion), Day 8 and Day 15
Population: PK samples were not analyzed as the study was terminated prematurely due to lack of operational feasibility and the halt of figitumumab development.
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Figitumumab
Time Frame: Cycle 2: Day 1 (within 2 hours before and 1 hour after figitumumab infusion); Cycle 3 to Cycle 17: Day 1 (within 2 hours before figitumumab infusion); end of treatment; 90-day follow-up visit
Population: as for outcome 4
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cycle 1: Plasma Concentration at the Last Quantifiable Time Point (Clast) of Figitumumab
Time Frame: Cycle 1: Day 1 (within 2 hours before figitumumab infusion), Day 2 (1 hour post figitumumab infusion), Day 8 and Day 15
Population: as for outcome 4
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Plasma Concentration at the Last Quantifiable Time Point (Clast) of Figitumumab
Description: Plasma Concentration at the Last Quantifiable Time Point (Clast) of Figitumumab from Cycle 2 to the end of treatment.
Time Frame: as for outcome 5
Population: as for outcome 4
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cycle 1: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Figitumumab
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) of figitumumab in cycle 1.
Time Frame: Days 1, 2, 8 and 15 of Cycle 1; Day 1 of subsequent cycle starting from Cycle 2 (up to Cycle 17); end of treatment ( 21 days after last dose of figitumumab); follow-up visit (90 days after last dose of figitumumab)
Population: as for outcome 4
Groups:
- Figitumumab 20 mg/kg + Pegvisomant 20 mg: Figitumumab 20 milligram/kilogram (mg/kg) intravenously over 1 to 2.5 hours on Day 1 and 2 of Cycle 1 and on Day 1 of subsequent cycles (up to total duration of 27 cycles). Pegvisomant 40 mg subcutaneously on Day 15 of Cycle 1 or Day 1 of Cycle 2 and thereafter pegvisomant 20 mg subcutaneously once daily up to total duration of 27 cycles. Each cycle was of 21 days.
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20 mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)of Figitumumab
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)of figitumumab after Cycle 1
Time Frame: as for outcome 5
Population: as for outcome 4
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Area Under the Trough Concentrations (AUCtrough)
Description: The trough concentration-time profile (AUCtrough) of pegvisomant was to be analyzed by noncompartmental methods.
Time Frame: Cycle 1: Day 15 (within 2 hours before loading dose), Day 16 (within 2 hours pre-SC dose); Cycle 2: Days 1, 8 and 15 (within 2 hours pre-SC dose); Cycle 3 up to Cycle 17: Day 1 (within 2 hours pre-SC dose); end of treatment; 90-day follow-up visit
Population: as for outcome 4
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean Change in Glucose Levels Between Fasting and Post Glucose Load
Description: The effect of combining figitumumab with pegvisomant was analyzed to assess whether pegvisomant reverses figitumumab-induced glucose intolerance at various pegvisomant dose levels. The change in glucose load was assessed by Glucose Tolerance Testing (GTT) at baseline (fasting), during Cycle 1 following administration of figitumumab alone (post load), and near the end of Cycle 2 (post load) following combined therapy with figitumumab and pegvisomant.
Time Frame: Screening; Day 8 of Cycle 1; Day 15 of Cycle 2
Population: Glucose tolerance set: All enrolled participants who started treatment and who had at least one baseline or on-study sample submitted. N=number of participants with analyable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 17 | 6
milligram/deciliter (mg/dL)
  Screening (n = 17, 6) | 30.35 (34.02) | 4.67 (17.60)
  Cycle 1 Day 8 (n = 15, 5) | 37.68 (30.95) | 15.40 (32.04)
  Cycle 2 Day 15 (n = 4, 5) | 55.15 (49.35) | 13.40 (28.35)

12. Secondary Outcome: Percentage of Participants Reporting Positive Anti-Drug Antibodies (ADA) Response for Figitumumab
Description: Percentage of participants with positive total or neutralizing ADA for figitumumab.
Time Frame: Day 1 of Cycles 1 and 4; end of treatment (21 days after last dose of figitumumab); follow-up visit (90 days after last dose of figitumumab)
Population: ADA samples were not analyzed as the study was terminated prematurely due to lack of operational feasibility and the halt of figitumumab development.
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST)version 1.1. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST version 1.1. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: From Screening, odd numbered cycles (predose, Cycle 3, 5, 7 etc.) up to Cycle 27 or end of treatment visit (21 days after last dose of figitumumab)
Population: Response-evaluable set: All participants who started Cycle 1 with an adequate baseline tumor assessment and at least 1 follow up tumor assessment.
Measure: Number; unit: participants
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20mg/kg + Pegvisomant 20 mg
Number analyzed (Participants) | 17 | 6
participants | 0 | 3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Figitumumab 20 mg/kg + Pegvisomant 10 mg | Figitumumab 20 mg/kg + Pegvisomant 20 mg
Serious Adverse Events (participants affected / at risk) | 9/17 | 4/6
Other Adverse Events (participants affected / at risk) | 17/17 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 20 mg/kg + Pegvisomant 10 mg (N=17) | Figitumumab 20 mg/kg + Pegvisomant 20 mg (N=6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 4 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 20 mg/kg + Pegvisomant 10 mg (N=17) | Figitumumab 20 mg/kg + Pegvisomant 20 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 2
Chills (General disorders) | 2 | 0
Disease progression (General disorders) | 2 | 0
Exercise tolerance decreased (General disorders) | 1 | 0
Fatigue (General disorders) | 13 | 4
General physical health deterioration (General disorders) | 0 | 1
Injection site induration (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Medical device pain (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Necrosis (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 2
Blood uric acid increased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 3 | 1
Insulin-like growth factor increased (Investigations) | 0 | 2
International normalised ratio increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 3 | 3
Weight increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0
Paraesthesia mucosal (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to lack of operational feasibility and the halt of figitumumab development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.